CLINICAL TRIAL: NCT03006523
Title: Impact of Inseminated Volume and Live Birth Rates After Intrauterine Insemination (IUI) With Donor Sperm (dIUI): A Prospective Randomized COntrolled Trial
Brief Title: 0.2 ml vs. 0.5 Inseminated Volume in Donor Intrauterine Insemination Cycles: A Prospective RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Jorge Rodriguez-Purata, Attending Physician of IVF Center, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMD-DEX-2016-03
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Infertility; Infertility, Male; Same-Sex Marriage; Parent, Single
Keywords: donor intrauterine insemination; insemination volume; Live Birth Rates; donor sperm
MeSH Terms: conditions — Infertility; Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrauterine Insemination with 200 µl (Active Comparator): The sperm sample will be concentrated by centrifugation to a volume of 200 µl
  Interventions: Procedure: Intrauterine insemination
- Intrauterine Insemination with 500 µl (Experimental): The sperm sample will be concentrated by centrifugation to a volume of 500 µl.
  Interventions: Procedure: Intrauterine insemination

INTERVENTIONS:
Procedure: Intrauterine insemination — IUI will be performed with a Wallace® insemination 2 Catheter (Cooper Surgical, Trumbull, CT, USA) depositing 0.2 or 0.5 ml of the sperm sample at the uterine fundus. All IUIs will be performed between 12 p.m. and 4 p.m. After the procedure, 10 min of bed rest will be prescribed. Inseminations will be performed every day of the week, including weekends.

SUMMARY:
To prospectively determine the most appropriate inseminated volume in donor IUI cycles. It is hypothesized that if the procedure is performed with 0.5 mL instead of 0.2, higher clinical pregnancy rates will be achieved by promoting higher sperm densities in the fallopian tubes at the time of ovulation by decreasing the amount of sperm cells lost during preparation and handling.

DETAILED DESCRIPTION:
A prospective RCT will be performed, including patients undergoing dIUI under ovulation induction. The trial is established to compare two inseminated volumes, 0.2 ml (control group) and 0.5 mL (study group), and will be conducted at the Reproductive Medicine Service of the Dexeus Women's Health Center. The Institutional Review Board has approved the research project and an informed consent will be obtained from all patients participating to the study.

All patients will undergo a full infertility investigation including hormonal evaluation between day 2 and day 5 of the cycle and confirmation of patency of the Fallopian tubes. Patients eligible for the study are between 18 and 40 years old, with regular menstrual cycles (21 - 35 days). Indications for the use of donor sperm are male factor infertility due to azoospermia or severe oligoasthenoteratozoospermia (requiring donor sperm), the presence of a heritable genetic disorder in the male partner, a single-parent request or same-sex couples' partners undergoing IUI. Exclusion criteria are the presence of tubal factor infertility, ≥grade III endometriosis, more than 3 previous dIUI cycles, or patients in whom ≥3 follicles >14mm are observed during the cycle. The randomization procedure will take place the day the donor IUI procedure. The randomization will be performed on the IUI cycle level. Randomization into one of the two groups will be performed using an open computer-generated list.

IUI will be performed with a Wallace® catheter depositing 0.2 or 0.5 ml of the sperm sample at the uterine fundus. All IUIs will be performed between 12 p.m. and 4 pm. After the procedure, 10 min of bed rest will be prescribed. Inseminations will be performed every day of the week, including weekends.

ELIGIBILITY:
Inclusion Criteria:

* All patients will undergo a full infertility investigation including hormonal evaluation between day 2 and day 5 of the cycle and confirmation of patency of the Fallopian tubes.
* Patients eligible for the study are between 18 and 40 years old and with regular menstrual cycles (21 - 35 days). Indications for the use of donor sperm are severe male factor infertility requiring donor sperm, the presence of a heritable genetic disorder in the male partner, a single-parent request or same-sex couples' partners undergoing IUI.
* Exclusion criteria are the presence of tubal factor infertility, grade III-IV endometriosis, more than 3 previous failed dIUI cycles, or patients in whom ≥3 follicles >14mm are observed during the IUI cycle. Patients will be included in the study only once. The randomization will be performed on the IUI cycle level. The group allocation will take place the day the dIUI and the biologist will randomized all included patients into one of the two groups using an open computer-generated list.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Ten months after insemination procedure

SECONDARY OUTCOMES:
Miscarriage rate | Any pregnancy loss before week 20
  Miscarriage was defined as a loss following a positive pregnancy test and/or detectable GS

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Rodriguez-Purata, MD, Principal Investigator — Fundacion Dexeus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veltman-Verhulst SM, Cohlen BJ, Hughes E, Heineman MJ. Intra-uterine insemination for unexplained subfertility. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD001838. doi: 10.1002/14651858.CD001838.pub4. PMID 22972053
- [Background] Cohlen BJ, Vandekerckhove P, te Velde ER, Habbema JD. Timed intercourse versus intra-uterine insemination with or without ovarian hyperstimulation for subfertility in men. Cochrane Database Syst Rev. 2000;(2):CD000360. doi: 10.1002/14651858.CD000360. PMID 10796711
- [Background] Goverde AJ, McDonnell J, Vermeiden JP, Schats R, Rutten FF, Schoemaker J. Intrauterine insemination or in-vitro fertilisation in idiopathic subfertility and male subfertility: a randomised trial and cost-effectiveness analysis. Lancet. 2000 Jan 1;355(9197):13-8. doi: 10.1016/S0140-6736(99)04002-7. PMID 10615885
- [Background] ESHRE Capri Workshop Group. Intrauterine insemination. Hum Reprod Update. 2009 May-Jun;15(3):265-77. doi: 10.1093/humupd/dmp003. Epub 2009 Feb 23. PMID 19240042
- [Derived] Rodriguez-Purata J, Latre L, Ballester M, Gonzalez-Llagostera C, Rodriguez I, Gonzalez-Foruria I, Buxaderas R, Martinez F, Barri PN, Coroleu B. Clinical success of IUI cycles with donor sperm is not affected by total inseminated volume: a RCT. Hum Reprod Open. 2018 Feb 15;2018(2):hoy002. doi: 10.1093/hropen/hoy002. eCollection 2018. PMID 30895244